CLINICAL TRIAL: NCT02066090
Title: Effects of Acupuncture on Serum Metabolic Parameters in Pre-menopausal Obese Women: A Randomized Controlled Trial
Brief Title: Acupuncture for Obesity on Serum Metabolic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Mi-Yeon Song, Professor, K.M.D., Ph.D., Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHNMCOH 2013-01-020
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Obesity
Keywords: acupuncture; obesity; metabolomics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real acupuncture (Experimental): manual acupuncture + electroacupuncture, twice a week, for 6 weeks
  Interventions: Device: Real acupuncture
- Sham acupuncture (Sham Comparator): sham acupuncture + placebo acupuncture without electrical stimulation, twice a week, for 6 weeks
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Real acupuncture — manual acupuncture (bilateral LI4, LI11, SP6, ST25, ST28, ST36) + electroacupuncture (middle CV6, CV12), twice a week, for 6 weeks
  common approaches for the treatment of obesity used by doctors of Korean medicine in Korea today
  Arms: Real acupuncture
Device: Sham acupuncture — sham acupuncture (bilateral LI4, LI11, SP6, ST25, ST28, ST36) + placebo acupuncture without electrical stimulation (middle CV6, CV12), twice a week, for 6 weeks
  sham acupuncture (0.25mm diameter x 40mm length, stainless steel, Acuprime, UK) as control for manual acupuncture (0.25mm diameter x 40mm length, stainless steel, Dongbangacupuncture Inc., Korea)
  placebo acupuncture without electrical stimulation as control for electroacupuncture (0.25mm diameter x 90mm length, stainless steel, Dongbangacupuncture Inc., Korea)
  Arms: Sham acupuncture

SUMMARY:
This research is planned to build a basis about the effect of acupuncture on serum metabolic parameters in pre-menopausal obese women with economic evaluation.

DETAILED DESCRIPTION:
It is consisted with two sub research.

First, clinical research to assess the effect of acupuncture for obesity on serum metabolic parameters will be processed with randomized, patient-assessor blinding, and sham-acupuncture controlled study design. 120 subjects would be collected and divided into two groups(experimental and placebo, 60 subjects each). Experimental group will undergo with real acupuncture treatment(manual acupuncture + electroacupuncture) twice a week, for 6 weeks. The effect on serum metabolic parameters will be assessed at 0 and 6 weeks.

Second is qualitative research to make a basis through the evaluation of economic efficacy and patients' satisfaction with acupuncture treatment for obesity.

ELIGIBILITY:
Inclusion Criteria:

* volunteers through announcements and advertisements
* premenopausal adult women (19 years of age or more)
* clinical diagnosis of obesity (Body mass index: 25 kg/m2 or more)

Exclusion Criteria:

* previously or currently having endocrine disease such as hypothyroidism or Cushing's syndrome, heart disease, lung disease, diabetes, malignant tumor, cholelithiasis, severe kidney impairment, severe liver impairment, anorexia nervosa or hyperorexia
* experience of taking medicines which might affect body weight and the concentration of serum metabolic parameters such as anorectic, laxative, oral steroid, thyroid hormone, amphetamine, cyproheptadine, phenothiazine, or medicines affecting absorption, metabolism, and excretion in the past 3 months
* experience of taking beta-blocker or diuretic for the treatment of hypertension in the past 3 months
* surgical treatment for the treatment of obesity
* currently or might be pregnant or breast-feeding
* experience of taking other experimental medicines in the past month
* weight loss of 10% or more of previous body weight in the past 6 months
* who stopped smoking in the past 3 months or who have irregular smoking habit
* pacemaker
* currently receiving any treatment for obesity
* other inadequate subjects assessed by the study investigators

Ages: 19 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
change in serum metabolic profile | before treatment at week1 (baseline) and after treatment at week6 (endpoint)

SECONDARY OUTCOMES:
change in body weight | baseline, 1, 2, 3, 4, 5, and 6 weeks
  using bioelectrical impedance analysis (BIA)
change in body fat mass | baseline, 1, 2, 3, 4, 5, and 6 weeks
  using bioelectrical impedance analysis (BIA)
change in muscle mass | baseline, 1, 2, 3, 4, 5, and 6 weeks
  using bioelectrical impedance analysis (BIA)
change in waist circumference | baseline, 1, 2, 3, 4, 5, and 6 weeks
change in hip circumference | baseline, 1, 2, 3, 4, 5, and 6 weeks
change in Beck Depression Index (BDI) | baseline and 6 weeks
change in Social Readjustment Rating Scale (SRRS) | baseline and 6 weeks
change in Stress Response Inventory (SRI) | baseline and 6 weeks
change in International Physical Activity Questionnaire (IPAQ) | baseline and 6 weeks
change in Fatigue Severity Scale (FSS) | baseline, 1, 2, 3, 4, 5, and 6 weeks
heart rate variability (HRV) | just before treatment at visit1(baseline), 10 minutes after treatment at visit1, just before treatment at visit12 (6 weeks), 10 minutes after treatment at visit12(end point)
number of participants with adverse events | up to the end of study
  * assessment of severity: mild, moderate, severe
  * assessment of relation: definitely related, probably related, possibly related, probably not related, definitely not related, unknown

OTHER OUTCOMES:
change in Measure Yourself Medical Outcome Profile (MYMOP) | baseline, 1, 2, 3, 4, 5, and 6 weeks
  outcome measure for the evaluation of patients' satisfaction and economic efficacy in secondary sub-study
change in EuroQol-5 Dimension (EQ-5D) | baseline and 6 weeks
  outcome measure for the evaluation of patients' satisfaction and economic efficacy in secondary sub-study

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Yeon Song, Ph.D., Principal Investigator — Department of Rehabilitation Medicine of Korean Medicine, Kyung Hee University Gangdong Hospital
Locations (1):
- Kyung Hee University Korean Medicine Hospital at Gangdong, Seoul, South Korea

REFERENCES:
- [Derived] Kim KW, Shin WC, Choi MS, Cho JH, Park HJ, Yoo HH, Song MY. Effects of acupuncture on anthropometric and serum metabolic parameters in premenopausal overweight and obese women: a randomized, patient- and assessor-blind, sham-controlled clinical trial. Acupunct Med. 2021 Feb;39(1):30-40. doi: 10.1177/0964528420912259. Epub 2020 Apr 17. PMID 32299241
- [Derived] Kim KW, Yoo HH, Cho JH, Yang YC, Kim JI, Kim SY, Park JY, Park HJ, Song MY. Effects of acupuncture on serum metabolic parameters in premenopausal obese women: study protocol for a randomized controlled trial. Trials. 2015 Aug 4;16:327. doi: 10.1186/s13063-015-0867-y. PMID 26238111